CLINICAL TRIAL: NCT06810427
Title: A Novel, Low-Cost, Handheld 3D Imaging System for Improved Screening for Cervical Neoplasia in Resource-Limited Settings
Acronym: CervImage
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pensievision, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB-24-2185; 2R44CA254586-02 (NIH)
Record Dates: First submitted 2025-01-25; First posted 2025-02-05 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Cervical Lesion; Intraepithelial dysplasia; Human Papillomavirus (HPV); CervImage
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Intervention Model Description: Single-center, pilot study of the CervImage [Pensievision, San Diego, CA] device utilizing an (1) human papillomavirus (HPV) or Intraepithelial dysplasia (CIN) group and (2) no-HPV/CIN group with a single study intervention [CervImage device] for collection of quantitative data regarding imaging quality over the standard-of-care imaging modality and qualitative feedback from physician and subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- CervImage Device (Experimental): CervImage device for cervical imaging to detect cervical intraepithelial dysplasia [CIN] via colposcopy
  Interventions: Device: CervImage device

INTERVENTIONS:
Device: CervImage device — CervImage™, developed by Pensievision, Inc., is an accessible, simple, cost-effective, early detection imaging technology for preventing cervical cancer deaths caused by a lack of screening.
  The novel device is a simple-to-operate, point-of-care, all-focus, 3D-imaging device, with clinical relevance to early-stage detection and prevention of cervical cancers. CervImage's proprietary 3D-rendering software, incorporating strategies previously used for high resolution imaging with NASA telescopes, can quantify tissue color, volume and shape. Virtual navigation tools and all-focus imaging enable straightforward use by minimally trained personnel; expert personnel can also benefit from shorter setup times.
  The research procedure and evaluation will be incorporated into the scheduled annual pap smear exam or colposcopic gynecologic exam that involves using a vaginal speculum.
  Other Names: CervImage

SUMMARY:
The purpose of this study is to evaluate the design and engineering of a new minimally invasive medical imaging device (CervImage™). Investigators are trying to find out if CervImage™ is reliable and easy to use to obtain clinical 3D photographs and to record 3D measurements in human cervixes. Investigators then plan to use these images to determine if CervImage™ design and engineering improvements need to be made.

DETAILED DESCRIPTION:
This study intends to evaluate the design and engineering of an innovative, minimally invasive, 3D, and medical imaging device (CervImage™) for detecting cervical lesions. The research procedure and evaluation will be incorporated into the scheduled annual pap smear exam or colposcopic gynecologic exam that involves using a vaginal speculum. The CervImage™ camera will be positioned within the speculum approximately 1-2 cm distal to the cervix. It will not come into physical contact with the participant. Data collection with the CervImage TM imaging device is expected to take less than 5 minutes. The study will generate live cervical images and gather qualitative feedback from both clinicians and participants. CervImage™ is not a diagnostic product, and this study will not be generating any efficacy or imaging data to be used for diagnostic or therapeutic purposes. If any abnormalities are observed in the CervImage™ procedure described, they will be further evaluated by the Principal Investigator. This will take place during the participant's routine gynecologic exam with colposcopy included as part of their scheduled clinical visit. The device will not be used for diagnostic purposes or for making any clinical decisions or recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Patient 21 to 70 years of age at screening
* Patients with known HPV infection or cervical intraepithelial neoplasia (16 patients)
* Healthy patients without history of HPV/CIN (2 patients)
* Participants able to consent for themselves

Exclusion Criteria:

* Cognitive Impairment
* Currently Pregnant
* Incarcerated Individual
* Any condition which in the clinical judgement of the PI makes the subject unsuitable or unsafe for study enrollment

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant must have cervix at time of study participation
Enrollment: 18 (Actual)
Dates: Start 2025-01-16 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-07-16 (Estimated)

PRIMARY OUTCOMES:
Image Quality and Resolution vs Standard-of-Care | Immediately after the procedure
  CervImage images evaluated on Spatial resolution, distortion, brightness, magnification, color correctness, corrupted pixel rows, and visual inspection vs standard-of-care cervical imaging for intraepithelial dysplasia [CIN] visualization.

SECONDARY OUTCOMES:
Time to Obtain Images | Immediately after the procedure
  Time required by the physician to obtain cervical images needed with the CervImage device vs standard-of-care device.
Comfort/Discomfort of Subject | Immediately after the procedure
  Subjective assessment of discomfort [and comfort] with using the CervImage device vs standard-of-care device for colposcopy, by the subject through use of a quantitative questionnaire with a scale of 1 to 10 with 1 being no pain and 10 being extremely painful.
Physician Satisfaction | Immediately after the procedure
  Overall satisfaction with use of the CervImage device vs standard-of-care device by physician using a quantitative questionnaire with a scale of 1 to 10 with 1 being dissatisfied and 10 being completely satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Isaiah Johnson, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Hull R, Mbele M, Makhafola T, Hicks C, Wang SM, Reis RM, Mehrotra R, Mkhize-Kwitshana Z, Kibiki G, Bates DO, Dlamini Z. Cervical cancer in low and middle-income countries. Oncol Lett. 2020 Sep;20(3):2058-2074. doi: 10.3892/ol.2020.11754. Epub 2020 Jun 19. PMID 32782524
- [Background] Gerstl S, Lee L, Nesbitt RC, Mambula C, Sugianto H, Phiri T, Kachingwe J, Llosa AE. Cervical cancer screening coverage and its related knowledge in southern Malawi. BMC Public Health. 2022 Feb 14;22(1):295. doi: 10.1186/s12889-022-12547-9. PMID 35164716
- [Background] Fuzzell LN, Perkins RB, Christy SM, Lake PW, Vadaparampil ST. Cervical cancer screening in the United States: Challenges and potential solutions for underscreened groups. Prev Med. 2021 Mar;144:106400. doi: 10.1016/j.ypmed.2020.106400. Epub 2021 Jan 1. PMID 33388330
- [Background] Suk R, Hong YR, Rajan SS, Xie Z, Zhu Y, Spencer JC. Assessment of US Preventive Services Task Force Guideline-Concordant Cervical Cancer Screening Rates and Reasons for Underscreening by Age, Race and Ethnicity, Sexual Orientation, Rurality, and Insurance, 2005 to 2019. JAMA Netw Open. 2022 Jan 4;5(1):e2143582. doi: 10.1001/jamanetworkopen.2021.43582. PMID 35040970
- [Background] Moucheraud C, Kawale P, Kafwafwa S, Bastani R, Hoffman RM. Health care workers' experiences with implementation of "screen and treat" for cervical cancer prevention in Malawi: A qualitative study. Implement Sci Commun. 2020 Dec 14;1(1):112. doi: 10.1186/s43058-020-00097-3. PMID 33317633
- [Background] Gupta R, Gupta S, Mehrotra R, Sodhani P. Cervical Cancer Screening in Resource-Constrained Countries: Current Status and Future Directions. Asian Pac J Cancer Prev. 2017 Jun 25;18(6):1461-1467. doi: 10.22034/APJCP.2017.18.6.1461. PMID 28669152
- [Background] Carson, J. C., Eikenberry, S. S., Smith, J. J. & Cordes, J. M. The Cornell High-Order Adaptive Optics Survey for Brown Dwarfs in Stellar Systems. II. Results from Monte Carlo Population Analyses. The Astronomical Journal 132, 1146 (2006). https://doi.org:10.1086/505705
- [Background] Carson, J. C. et al. A DISTANCE-LIMITED IMAGING SURVEY OF SUBSTELLAR COMPANIONS TO SOLAR NEIGHBORHOOD STARS. The Astronomical Journal 137, 218 (2009).
- [Background] Durkan, S., Janson, M. & Carson, J. C. HIGH CONTRAST IMAGING WITH SPITZER: CONSTRAINING THE FREQUENCY OF GIANT PLANETS OUT TO 1000 au SEPARATIONS. The Astrophysical Journal 824, 58 (2016). https://doi.org:10.3847/0004-637X/824/1/58
- [Background] Carson, J. C. et al. A SPITZER IRAC IMAGING SURVEY FOR T DWARF COMPANIONS AROUND M, L, AND T DWARFS: OBSERVATIONS, RESULTS, AND MONTE CARLO POPULATION ANALYSES. The Astrophysical Journal 743, 141 (2011). https://doi.org:10.1088/0004-637X/743/2/141
- [Background] Carson, J. et al. DIRECT IMAGING DISCOVERY OF A "SUPER-JUPITER" AROUND THE LATE BTYPE STAR κ And*. The Astrophysical Journal Letters 763, L32 (2013). https://doi.org:10.1088/2041- 8205/763/2/L32
- [Background] Carson, B., Carson, J., Esener, S. & Liu, K. U.S. Provisional Patent: Method, System, Software and Device for Remote, Miniaturized, and Three- Dimensional Imaging and Analysis of Human Lesions; Research and Clinical Applications. (2019).
- [Background] Baghdadchi S, Liu K, Knapp J, Prager G, Graves S, Akrami K, Manuel R, Bastos R, Reid E, Carson D, Esener S, Carson J, Liu YT. An innovative system for 3D clinical photography in the resource-limited settings. J Transl Med. 2014 Jun 15;12:169. doi: 10.1186/1479-5876-12-169. PMID 24929434
- [Background] WHO Guidelines for Screening and Treatment of Precancerous Lesions for Cervical Cancer Prevention. Geneva: World Health Organization; 2013. Available from http://www.ncbi.nlm.nih.gov/books/NBK195239/ PMID 24716265
- [Background] Byun JM, Kim YN, Jeong DH, Kim KT, Sung MS, Lee KB. Three-dimensional transvaginal ultrasonography for locally advanced cervical cancer. Int J Gynecol Cancer. 2013 Oct;23(8):1459-64. doi: 10.1097/IGC.0b013e3182a16997. PMID 24257560
- See also: Pensievision, Inc - CervImage — https://www.pensievision.com/

DOCUMENTS (1):
  • Informed Consent Form (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT06810427/ICF_000.pdf